CLINICAL TRIAL: NCT05188209
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG003 in EGFR-Positive, HER2-Negative Advanced Gastric Cancer.
Brief Title: A Study to Evaluate the Efficacy and Safety of MRG003 in Patients With Advanced Gastric Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-006
Record Dates: First submitted 2022-01-05; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Advanced or Metastatic Gastric Cancer; Advanced or Metastatic Gastroesophageal Junction Carcinoma
Keywords: MRG003; Antibody Drug Conjugate (ADC); Gastric Cancer; EGFR-positive, HER2-negative
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003 (Experimental): On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.0 mg/kg calculated based on the actual body weight
  Interventions: Drug: MRG003

INTERVENTIONS:
Drug: MRG003 — Administered intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG003 in patients with EGFR-positive, HER2-negative, inoperable locally advanced or metastatic gastric cancer.

DETAILED DESCRIPTION:
Approximately 6054 patients will be enrolled to evaluate the safety and preliminarily efficacy of MRG003. Patients will receive 2.0 mg/kg dose of MRG003 intravenously every 3 weeks (Q3W) and may receive up to 24 months of MRG003 if there is evidence of clinical benefit to the patients.

ELIGIBILITY:
Inclusion Criteria:

* - Willing to sign the ICF and follow the requirements specified in the protocol.
* Age: 18-75 years (including 18 and 75), both genders.
* Expected survival time≥3 months.
* Patients with histologically confirmed inoperable locally advanced or metastatic gastric adenocarcinoma.
* Tumor tissue must be EGFR positive and HER2 negative.
* Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* ECOG performance score 0 or 1.
* Organ functions and coagulation function must meet the basic requirements.
* No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%.
* Serum or urine pregnancy test negative within 7 days before the first dose of investigational drug.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* - Squamous cell carcinoma, carcinoid, neuroendocrine carcinoma, undifferentiated carcinoma, or other gastric cancers,or adenocarcinoma with other pathological components that cannot be classified, or adenocarcin oma accompanied by other pathological components.
* History of hypersensitivity to any component of the study drug or to other EGFR-targeting agents.
* Antitumor biological therapy or immunotherapy, targeted small molecule therapy and have history of systemic chemotherapy within 4 weeks before the first administration of the investigational drug, or major surgery. Traditional Chinese medicine, Chinese patent medicine or traditional Chinese medicine formula with anti-tumor effect should not be used within 2 weeks before the first administration.
* Potent CYP3A4 inhibitors or inducers are in use and cannot be discontinued.
* Known active CNS metastasis.
* Uncontrolled pleural effusion, pericardial effusion or recurrent ascites.
* Patients with intestinal obstruction requiring treatment were excluded.
* Residual toxicity reactions caused by previous anti-tumor treatment or abnormal values of laboratory tests higher than grade 1 (CTCAE v5.0).

Peripheral neuropathy ≥ Grade 2 (NCICTCAE version 5.0).

* Uncontrolled or poorly controlled hypertension.
* Uncontrolled or poorly controlled heart disease.
* Known active hepatitis B or C.
* Active bacterial, viral, fungal, rickettsia, or parasitic infections that require systemic anti-infective treatment.
* Known history of malignancy.
* History of ophthalmologic abnormalities
* History of severe skin disease
* Moderate to severe dyspnea at rest caused by advanced cancer or its complications, or severe primary lung disease, oxygen saturation < 93% in non-oxygen state, or history of any interstitial lung disease or interstitial lung disease (ILD) requiring oral or intravenous glucocorticoids or non-infectious pneumonia.
* Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy.
* History of pulmonary embolism or deep vein thrombosis within 6 months before the first administration of the investigational drug.
* Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy.

Decompensated cirrhosis of Child-Pugh class B, C

* Complicated with severe, uncontrolled infection or known human immunodeficiency virus (HIV) infection, or diagnosed as acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or history of allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or solid organ transplantation.
* Vaccination of live virus vaccine within 30 days before the first administration of the study drug. Inactivated seasonal influenza vaccine or approved COVID-19 vaccine is allowed.
* Uncontrolled intercurrent illness
* Patients requiring parenteral nutrition within 4 weeks
* Women who are lactating or pregnant.
* Other conditions that in the clinical judgement of the investigator make the patient not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-03-21 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by Independent Review Committee (IRC) according to RECIST v1.1.
Adverse Events (AEs) | Baseline to 30(for AE) and 45(for SAE) days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Duration of Response (DoR) | Baseline to study completion (up to 24 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportions of patients achieving CR, PR, and stable disease (SD) after treatment.
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.
PK parameter for MRG003: (Cmax) | Baseline to 30 days after the last dose of study treatment
  Maximum observed plasma concentration.
PK parameter for MRG003: (AUClast) | Baseline to 30 days after the last dose of study treatment
  Area under the curve up to the last validated measurable plasma concentration
PK parameter for total antibody (TAb): Cmax | Baseline to 30 days after the last dose of study treatment
  Maximum observed plasma concentration.
PK parameter for TAb: AUClast | Baseline to 30 days after the last dose of study treatment
  Area under the curve up to the last validated measurable plasma concentration
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Baseline to 30 days after the last dose of study treatment
  Maximum observed plasma concentration.
PK parameter for MMAE: AUClast | Baseline to 30 days after the last dose of study treatment
  Area under the curve up to the last validated measurable plasma concentration
The proportion of patients with positive of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No